CLINICAL TRIAL: NCT04550754
Title: Evaluation of the Medical Management of Tramadol Use Disorders in Patients Hospitalized for Tramadol Withdrawal
Brief Title: Evaluation of the Management of Tramadol Use Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0430
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Withdrawal
Keywords: Substance use disorder; Programme de Medicalisation des Systèmes d'Information; tramadol
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for tramadol withdrawal: Patients hospitalized for tramadol withdrawal in Montpellier University Hospital and Nîmes University Hospital from 01/01/2015 to 31/12/2019

SUMMARY:
In France, In recent years, there has been a steady increase in reports of abuse and dependence on tramadol. Over 50% of tramadol withdrawal syndromes involve taking tramadol in therapeutic doses, sometimes for short periods of less than a week. Physical dependence can develop when a therapeutic maintenance dose is prescribed for the treatment of mild to moderate pain. Due to its mixed mechanism of action, tramadol withdrawal syndromes are not only characterized by classic signs of opioid withdrawal (muscle pain, mydriasis, sweating, nausea and vomiting, tearing, rhinorrhea, yawning, fever, insomnia, etc.). The properties of this substance on serotonin explain the effects which are added to the morphine-mimetic withdrawal of tramadol. Analysis of spontaneous reports shows "psychological and psychic" signs of withdrawal. Currently, there is no validated protocol for the management of tramadol withdrawal. The main objective is to assess the different options for managing tramadol withdrawal: opioid maintenance therapy and symptomatic treatments, in relation to the addictive and psychiatric co-morbidities in patients. The study also provides insight into the different types of withdrawal syndromes experienced by patients in order to raise awareness among doctors when prescribing tramadol.

ELIGIBILITY:
Inclusion criteria:

* >18 years old
* Tramadol actual misuse/addiction
* Patients hospitalized for Tramadol withdrawal

Exclusion criteria:

* <18 years old
* History of misuse or addiction for tramadol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized in Montpellier University Hospital and Nîmes University Hospital for Tramadol withdrawal
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Medical Management of Tramadol withdrawal syndrome | 1 day
  Management by substitution drugs, by therapeutic degrowth

SECONDARY OUTCOMES:
Tramadol withdrawal syndrome experienced by patients | 1 day
  Description of classic cpioid withdrawal symptoms and atypical aymptoms apecific to

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Peyrière, PH, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC